CLINICAL TRIAL: NCT04629508
Title: A 2-Part, Phase 2, Open-Label Study of the Safety, Tolerability, and Efficacy of Itacitinib Immediate Release in Participants With Primary Myelofibrosis or Secondary Myelofibrosis (Post-Polycythemia Vera Myelofibrosis or Post-Essential Thrombocythemia Myelofibrosis) Who Have Received Prior Ruxolitinib and/or Fedratinib Monotherapy
Brief Title: To Assess the Safety, Tolerability and Efficacy of Itacitinib Immediate Release Tablets in Participants With Primary or Secondary Myelofibrosis Who Have Received Prior Ruxolitinib and/or Fedratinib Monotherapy (LIMBER-213)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB 39110-213/LIMBER-213; 2020-003123-42 (EudraCT Number); NCT04821791 (obsolete NCT alias)
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Myelofibrosis; Polycythemia Vera; Thrombocythemia
Keywords: Myelofibrosis; Post-PV Myelofibrosis; Post-ET Myelofibrosis; LIMBER; LIMBER-213; MF; Myeloproliferative Neoplasms
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera; Thrombocytosis; Myeloproliferative Disorders | interventions — itacitinib; INCB039110

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 : Dose Escalation of itacitinib (Experimental): Participants will be dosed at different dose levels with a maximum of up to 9 participants per dose level.
  Interventions: Drug: itacitinib
- Part 2 : Dose Expansion of itacitinib (Experimental): Participants will be dosed at the recommended Phase 2 dose (RP2D) identified in Part 1.
  Interventions: Drug: itacitinib

INTERVENTIONS:
Drug: itacitinib — itacitinb Immediate Release (IR) will be dosed orally twice a day
  Other Names: INCB039110

SUMMARY:
This is a 2-part study. In Part 1, participants will be dosed at 2 different dose levels in order to select the RP2D for Part 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary MF meeting the 2016 WHO criteria for overt PMF or secondary MF (PPV-MF or PET-MF) meeting the 2008 IWG-MRT criteria.
* At least Intermediate 1 risk MF according to the DIPSS.
* Prior treatment with ruxolitinib and/or fedratinib monotherapy
* Currently receiving ruxolitinib or fedratinib monotherapy for PMF or secondary MF.
* Splenomegaly defined as palpable spleen at least 5 cm below the left costal margin or volume ≥ 450 cm3 on imaging assessed during screening.
* Allogeneic stem cell transplant not planned.
* Platelet is greater than or equal to 50 × 109/L at screening.
* Ability to comprehend and willingness to sign a written ICF for the study.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Prior treatment with a JAK inhibitor other than ruxolitinib or fedratinib
* Record of ≥ 10% myeloid blasts in the peripheral blood (on peripheral blood smear) or bone marrow prior to or at the time of screening
* For participants on ruxolitinib or fedratinib, unable to be tapered from that treatment over the course of 14 days without corticosteroids, hydroxyurea, or other agents
* Treatment with ruxolitinib, fedratinib or other MF-directed therapy (approved or investigational) within 2 weeks of Day 1
* Prior splenectomy or splenic irradiation within 6 months before receiving the first dose of itacitinib
* Unable or unwilling to undergo serial MRI or CT scans for spleen volume measurement
* Unable or unwilling to complete MFSAF v4.0 diary on a daily basis during the study
* ECOG performance status ≥ 3
* Life expectancy less than 24 weeks
* Not willing to receive RBC or platelet transfusions
* Participants with laboratory values at screening outside of protocol defined ranges
* Significant concurrent, uncontrolled medical condition
* Participants with impaired cardiac function or clinically significant cardiac disease unless approved by medical monitor/sponsor
* History or presence of an abnormal ECG that, in the investigator's opinion, is clinically meaningful
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment.
* Evidence of HBV or HCV infection or risk of reactivation
* Known HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (8):
  - Tulane University, New Orleans, Louisiana
  - Rcca Md, Llc, Bethesda, Maryland
  - Midamerica Cancer Care, Kansas City, Missouri
  - New Jersey Hematology Oncology Associates Llc, Brick, New Jersey
  - Baptist Cancer Center, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Texas Oncology - Baylor Sammons Cancer Center, Dallas, Texas
  - Renovatio Clinical Consultants Llc, Spring, Texas
- Interne 1 - Hematologie Mit Stammzelltransplantation, Hemostaseologie Und Medizinische Onkologie Ord, Linz, Austria
- Belgium (4):
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Jessa Ziekenhuis, Hasselt
  - AZ DELTA, Roeselare
  - Chu Ucl Namur University Hospital Mont-Godinne, Yvoir
- Germany (2):
  - Universitaetsmedizin Greifswald, Greifswald
  - Universitatsklinikum Halle (Saale), Halle
- Italy (3):
  - Istituto Di Ricovero E Cura A Carattere Scientifico (Irccs) Ospedale San Raffaele, Milan
  - Aou San Giovanni Di Dio E Ruggi, Salerno
  - Treviso Hospital, Treviso
- Pratia Hematologia Katowice, Katowice, Poland
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari I Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: Related Info — https://www.incyteclinicaltrials.com/limber/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 3 study centers in the United States and Italy.
Groups:
- Itacitinib 300 mg: Participants received itacitinib immediate release 300 milligrams (mg) twice a day (BID) orally (PO) for at least 24 weeks. Participants could remain on treatment as long as they were receiving clinical benefit and had not met any criteria for treatment discontinuation.
Period: Overall Study
Arm/Group | Itacitinib 300 mg
Started | 4
Completed | 0
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Death | 2
Not completed — Protocol-specified withdrawal criterion met | 1

BASELINE CHARACTERISTICS:
Arm/Group | Itacitinib 300 mg
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug-related. An AE could therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE was defined as an AE that was reported for the first time or the worsening of a pre-existing event after the first dose of study treatment.
Time Frame: up to 724 days
Population: Safety Evaluable Population: all participants enrolled in the study who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Itacitinib 300 mg
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Part 1: Number of Participants With Any Grade 3 or Higher TEAE
Description: A TEAE was defined as an AE that was reported for the first time or the worsening of a pre-existing event after the first dose of study treatment. The severity of AEs was assessed using Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grades 1 through 5. The investigator made an assessment of intensity for each AE and SAE reported during the study and assigned it to 1 of the following categories: Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: up to 724 days
Population: Safety Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Itacitinib 300 mg
Number analyzed (Participants) | 4
Participants | 4

3. Primary Outcome: Part 2: Splenic Response Rate (SRR) at Week 24
Description: SRR was defined as the percentage of participants who had a reduction in spleen volume (by imaging) of at least 35% when compared with Baseline.
Time Frame: Baseline; Week 24
Population: Analysis was not conducted because Part 2 never opened for enrollment.
Arm/Group | Itacitinib 300 mg
Number analyzed (Participants) | 0

4. Secondary Outcome: Part 2: Number of Participants With Any TEAE
Description: as for outcome 1
Time Frame: up to at least 24 weeks
Population: Analysis was not conducted because Part 2 never opened for enrollment.
Arm/Group | Itacitinib 300 mg
Number analyzed (Participants) | 0

5. Secondary Outcome: Part 2: Number of Participants With Any Grade 3 or Higher TEAE
Description: as for outcome 2
Time Frame: up to at least 24 weeks
Population: Analysis was not conducted because Part 2 never opened for enrollment.
Arm/Group | Itacitinib 300 mg
Number analyzed (Participants) | 0

6. Secondary Outcome: Part 2: Total Symptom Score (TSS) Response Rate at Week 24
Description: TSS response was defined as the percentage of participants who achieved at least 50% reduction in TSS over the 28 days immediately before the end of Week 24 compared with the 7 days immediately before the initiation of itacitinib immediate release (aseline).B
Time Frame: Baseline; Week 24
Population: Analysis was not conducted because Part 2 never opened for enrollment.
Arm/Group | Itacitinib 300 mg
Number analyzed (Participants) | 0

7. Secondary Outcome: Part 2: Mean Change (From Day 1 Versus Week 12 and Week 24) in the 5 Multi-item Functional Scale Scores and the Multi-item Global Health Status Scale Score (EORTC QLQ-C30)
Description: The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) was to be used to assess the improvement in quality of life.
Time Frame: Baseline; Weeks 12 and 24
Population: Analysis was not conducted because Part 2 never opened for enrollment.
Arm/Group | Itacitinib 300 mg
Number analyzed (Participants) | 0

8. Secondary Outcome: Part 2: Percentage of Participants Categorized as Improved on the Week 24 Patient Global Impression of Change (PGIC)
Description: The PGIC consists of a single question pertaining to a participant's overall status since the start of the study. The questionnaire gives participants 7 options to describe their overall status including: very much improved, much improved, minimally improved, no change, minimally worse, much worse, and very much worse.
Time Frame: Baseline; Week 24
Population: Analysis was not conducted because Part 2 never opened for enrollment.
Arm/Group | Itacitinib 300 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 724 days
Description: Treatment-emergent adverse events (TEAEs), defined as AEs that were reported for the first time or the worsening of pre-existing events after the first dose of study treatment, were reported for the Safety Evaluable Population.
Groups:
- Itacitinib 300 mg: itacitinib 300 mg
- Total: Total
Arm/Group | Itacitinib 300 mg | Total
All-Cause Mortality (participants affected / at risk) | 2/4 | 2/4
Serious Adverse Events (participants affected / at risk) | 3/4 | 3/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Itacitinib 300 mg (N=4) | Total (N=4)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cytokine storm (Immune system disorders) | 1 (2) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Itacitinib 300 mg (N=4) | Total (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 2 (2) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 2 (4) | 2 (4)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The sponsor terminated study enrollment following an assessment regarding the expected duration of recruitment for the Phase 2 portion of the study combined with the availability of other study options for this patient population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT04629508/Prot_SAP_000.pdf